CLINICAL TRIAL: NCT05782062
Title: Pharmacomechanical Dialysis Access Salvage With Balloon Assisted Maceration Versus Rotational Thrombectomy
Brief Title: Balloon Assisted Maceration Versus Rotational Thrombectomy in Dialysis Access Salvage
Acronym: BART
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: funding
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Argon Medical Devices (Industry)
Responsible Party: Principal Investigator, Junaid Yasin Raja, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300010783
Record Dates: First submitted 2023-03-12; First posted 2023-03-23 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Dialysis Access Malfunction; Dialysis; Complications
Keywords: Thrombosis of dialysis access

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Rotational Thrombectomy (Experimental): Use of the Cleaner XT
  Interventions: Device: Cleaner XT
- Balloon Assisted maceration (Active Comparator): Use of angioplasty balloons for balloon maceration
  Interventions: Device: Balloon

INTERVENTIONS:
Device: Cleaner XT — Wire like device that rotates to allow for wall to wall disruption of thrombus.
  Arms: Rotational Thrombectomy
Device: Balloon — Use of balloon for disrupting thrombus.
  Arms: Balloon Assisted maceration

SUMMARY:
The purpose of this research study is to compare how well a wire like device disrupts and removes blood clot in your blocked dialysis graft/fistula in comparison to inflating a balloon in your access for the same purpose. The wire like device is called the Cleaner XT and has already been approved by the government/Food and Drug Administration (FDA) for this purpose.

Blood clots in your dialysis access can be fairly common and prevent you from being able to get dialysis. Procedures for opening this blockage must then be performed which is why you have been sent to the hospital today. There are different ways of opening up this blockage which can including blowing up a balloon in multiple areas of the graft/fistula to squeeze the blood clot to break up the blockage or using a wire like device to break up the clot in small pieces and try to remove all of the clot from the wall of the graft/fistula.

ELIGIBILITY:
Inclusion Criteria:

* End stage renal disease on hemodialysis
* Age greater than 18
* Upper extremity dialysis graft/fistula

Exclusion Criteria:

* Pregnant
* Incarcerated
* Age under 18
* Inability to consent for self
* Graft/fistula in a location other than upper extremity
* Peritoneal dialysis
* Catheter dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-15 (Estimated); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Secondary patency | 6 months post procedurally
  How long the dialysis access remains functional after the procedure.